CLINICAL TRIAL: NCT06935357
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Felzartamab in Adults With IgA Nephropathy (PREVAIL)
Brief Title: A Study to Learn About the Effects of Felzartamab Infusions on Adults With Immunoglobulin A Nephropathy (IgAN)
Acronym: PREVAIL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Human Immunology Biosciences, Inc. (HI-Bio) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 299IG301; 2024-519345-30-00 (Other: EU CT Number)
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Immunoglobulin A Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — felzartamab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants will receive several intravenous (IV) doses of felzartamab.
  Interventions: Drug: Felzartamab
- Cohort 2 (Placebo Comparator): Participants will receive several IV doses of placebo.
  Interventions: Drug: Placebo
- Cohort 3 (Experimental): Participants with an estimated glomerular filtration rate (eGFR) ≥ 20 and <30 milliliter per minute per 1.73 square meter (mL/min/1.73m^2) will receive several IV doses of felzartamab.
  Interventions: Drug: Felzartamab
- Cohort 4 (Placebo Comparator): Participants with an eGFR ≥ 20 and <30 mL/min/1.73m^2 will receive several IV doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Felzartamab — Administered IV
  Other Names: MOR202, MOR03087, TJ202, HIB202, BIIB148
  Arms: Cohort 1; Cohort 3
Drug: Placebo — Administered IV
  Arms: Cohort 2; Cohort 4

SUMMARY:
In this study, researchers will learn more about the use of felzartamab in participants with immunoglobulin A nephropathy (IgAN). This study will focus on participants who have protein in their urine (proteinuria) as a result of damaged kidneys.

The main goal of the study is to learn about the effect felzartamab has on proteinuria. The main question that researchers want to answer is:

• How much does the amount of protein in the urine change from the start of the study to Week 36?

Researchers will learn about the effect felzartamab has on the kidneys' ability to filter blood. They will also learn more about the safety of felzartamab and how it is processed by the body.

The study will be done as follows:

* Participants will be screened to check if they can join the study.
* Participants will be randomized to receive either felzartamab or a placebo. A placebo looks like the study drug but contains no real medicine.
* Neither the researchers nor the participants will know what the participants will receive.
* Participants will receive felzartamab or placebo as intravenous (IV) infusions. The treatment period will last 24 weeks.
* Afterwards, participants will enter a follow-up period which will last 80 weeks.
* In total, participants will have 17 study visits. Participants will stay in the study for about 2 years.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy of felzartamab compared to placebo on proteinuria in participants with Immunoglobulin A nephropathy (IgAN). The main secondary objective of the study is to evaluate the efficacy of felzartamab compared to placebo on kidney functions in participants with IgAN. The additional secondary objectives are to evaluate the efficacy of felzartamab compared to placebo on additional clinical endpoints and to assess the pharmacokinetics (PK) and immunogenicity of felzartamab.

ELIGIBILITY:
Key Inclusion Criteria:

* Biopsy-confirmed diagnosis of IgAN within the past 10 years prior to signature of the informed consent form (ICF). For participants with diabetes mellitus type 2, biopsy confirmation of IgAN diagnosis must be done within the past 24 months prior to signing the ICF.
* An eGFR ≥ 30 mL/min/1.73m^2 at Screening as calculated using the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine formula. An eGFR of ≥ 20 and < 30 mL/min/1.73m^2 is acceptable for the cohorts 3 and 4.
* Proteinuria of ≥ 1.0 gram per day (g/day) or UPCR ≥0.8 gram per gram (g/g) as assessed by an adequate 24-hour urine collection.
* Clinically stable on a maximally tolerated dose or maximally approved dose of angiotensin-converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) for at least 12 weeks prior to Screening, or intolerant of ACEI or ARB. If intolerant, this must be discussed with the Medical Monitor prior to randomization. Participants may also be using sodium-glucose cotransporter-2 inhibitors (SGLT2is), endothelin receptor antagonists (ERAs) approved for the treatment of IgAN, dual endothelin angiotensin receptor antagonist (DEARAs) approved for the treatment of IgAN, and/or mineralocorticoid receptor antagonists (MRAs) as long as the dose is stable for at least 12 weeks prior to Screening. Participants should remain on stable doses of these background medications for the duration of the study. Once the ICF is signed and thereafter, the doses cannot be changed during the study nor the drugs discontinued except if deemed related to an AE. Participants using sparsentan will not be permitted to use simultaneous ACEI or ARB medication.

Key Exclusion Criteria:

* Secondary forms of IgAN, indicated by the presence of any other systemic disease potentially leading to IgA deposits as determined by the Investigator.
* History of rapidly progressive variant of IgAN, defined as eGFR loss by > 50% per 3 months and not explained by changes in renin-angiotensin system (RAS) blockade or other factors.
* Nephrotic syndrome presumed to be due to minimal change disease (MCD) variant.
* Concomitant other progressive glomerulonephritis or non-immunologic glomerular disease such as diabetic nephropathy.
* Type 2 diabetes mellitus with Hemoglobin A1c (HbA1c) > 8% at Screening, or evidence of diabetic nephropathy on biopsy, history of diabetic microvascular or macrovascular disease (eg, diabetic retinopathy, peripheral neuropathy).
* Any diagnosed or suspected immunosuppressed or immunodeficient state such as asplenia, human immunodeficiency virus (HIV), primary immunodeficiencies, organ or bone marrow transplantation, with the exception of corneal transplants.
* Previously treated with immunosuppressive or other immunomodulatory agents such as but not limited to cyclophosphamide, rituximab, infliximab, eculizumab, canakinumab, mycophenolate mofetil (MMF) or mycophenolate sodium (MPS), cyclosporine, tacrolimus, sirolimus, everolimus, or systemic corticosteroids exposure (> 7.5 milligrams per deciliter [mg/d] prednisone/prednisolone equivalent) within 4 months (or 12 months for rituximab) prior to Screening.
* Participants currently treated with oral budesonide. Participants who have stopped this therapy ≥ 4 months prior to Screening may be eligible.
* Active clinically significant infections, known history of recurrent clinically significant infection, or Screening laboratory evidence consistent with an active infection, or IV anti-infectives (antibacterials, antiviral or antifungals). Participants with a history of opportunistic infections are excluded.
* Hypogammaglobulinemia: Serum Immunoglobin G (IgG) < 6.0 gram per litre (g/L), at Screening.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-06-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Proteinuria as Measured by the Urine Protein: Creatinine Ratio (UPCR) | Baseline up to Week 36

SECONDARY OUTCOMES:
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) Values Calculated Using the Chronic Kidney Disease Epidemiology (CKD-EPI) Creatinine Equation | Baseline up to Week 104
Percentage of Participants Achieving Complete Response (CR) | Baseline up to Week 104
  CR is defined as a UPCR value (based on 24-hour urine collection) of < 0.5 gram per gram (g/g), a reduction in UPCR of ≥ 50%, and a stable eGFR (decrease from baseline in eGFR of ≤ 25%).
Percentage of Participants who Progressed to Kidney Malfunction | Baseline up to Week 104
  The percentage of participants progressing to kidney malfunction will be reported based on one of the following, 1. ≥ 40% Reduction in eGFR Sustained for ≥ 30 Days, 2. eGFR <15 mL/min/1.73m^2 for ≥ 30 Days, 3. Undergoing Dialysis for ≥ 30 Days, 4. Undergoing Kidney Transplantation, 5. Died From Kidney Failure
Percentage of Participants Requiring Rescue Therapy | Baseline up to Week 104
Change From Baseline in eGFR Values Calculated Using the CKD-EPI Creatinine Equation | Baseline up to Week 52
Felzartamab Serum Concentrations Over Time | Predose and at multiple timepoints postdose up to Week 36
Number of Participants with Anti-Drug Antibodies (ADAs) Against Felzartamab | Baseline up to Week 104
Percentage of Participants With Treatment Emergent Adverse Event (TEAE) and Treatment Emergent Serious Adverse Event (TESAE) | Baseline up to Week 104
Number of Participants With Clinically Significant Change From Baseline in Vital Signs Abnormalities | Baseline up to Week 104
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to Week 104
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Abnormalities | Baseline up to Week 104
Number of Participants With Clinically Significant Change From Baseline in Physical Examinations Abnormalities | Baseline up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (190):
- United States (22):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Kidney & Hypertension Center - Apple Valley, Apple Valley, California
  - Scripps Green Hospital, Carlsbad, California
  - National Institute of clinical Research Administration Office, Garden Grove, California
  - FOMAT Medical Research - FOMAT - PPDS, Oxnard, California
  - North America Research Institute-San Dimas, San Dimas, California
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Royal Research, Corp., Hollywood, Florida
  - Central Florida Kidney Specialists, Orlando, Florida
  - CDC Research Institute, LLC, Port Saint Lucie, Florida
  - American Clinical Trials LLC, Acworth, Georgia
  - The Vasculitis and Glomerulonephritis Center at Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Elixia Health - Michigan Kidney Consultants, LLC - Elixia - PPDS, Pontiac, Michigan
  - Anointed Nephrology and HTN - SKYCRNG - PPDS, Brookhaven, Mississippi
  - Midwest Nephrology Associates,Inc., City of Saint Peters, Missouri
  - James J Peters Veterans Administration Medical Center - NAVREF - PPDS, The Bronx, New York
  - Lifespan at Rhode Island Hospital, Providence, Rhode Island
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Texas Kidney Institute - Dallas, Dallas, Texas
  - Provecta Research Network, Houston, Texas
  - R & H Clinical Research, Katy, Texas
- Argentina (5):
  - Hospital Italiano de Buenos Aires, Almagro, Ciudad Autónoma de BuenosAires
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - CIMER-Centro Integral de Medicina Respiratoria, San Miguel de Tucumán, Tucumán Province
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar - PPDS, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires
- Australia (4):
  - John Hunter Hospital, New Lambton, New South Wales
  - Concord Repatriation General Hospital, New South Wales, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Townsville Hospital, Douglas, Queensland
- Belgium (6):
  - Hôpital Erasme - PPDS, Anderlecht, Brussels Capital
  - ZOL Genk - campus Sint-Jan, Genk, Limburg
  - UZ Leuven - PPDS, Leuven, Vlaams Brabant
  - Jan Yperman, Ieper, West-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
- Brazil (7):
  - Freire Pesquisa Clínica, Belo Horizonte, Minas Gerais
  - Irmandade da Santa Casa de Misericórdia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Centro Mineiro de Pesquisa - CMiP, Juiz de Fora, Minas Gerais
  - Fundação Universidade de Caxias do Sul - Instituto de Pesquisas em Saúde, Caxias do Sul, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz- HAOC, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Bulgaria (4):
  - Medical Center Medconsult Pleven - Lovech Branch, Lovech
  - Medical Center Hera EOOD, Montana - Hera Clinics - PPDS, Montana
  - Medical Center Medconsult Pleven OOD, Pleven
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD-15 Acad. Ivan Geshov Blvd, Sofia
- McGill University Health Centre (MUHC), Montreal, Quebec, Canada
- China (27):
  - Fu Yang People's Hospital - South Campus, Fuyang, Anhui
  - The First Affiliated Hospital of Anhui Medical University - Jixilu Campus, Hefei, Anhui
  - Peking University First Hospital - Changqiao Campus, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University - Yanjiang Campus, Guangzhou, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Second Hospital of Hebei Medical University - Main, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Henan Science and Technology University - Jinghua Campus, Luoyang, Henan
  - Yichang Central People's Hospital - Wujiagang Campus, Yichang, Hubei
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai General Hospital - North Campus, Shanghai, Shanghai Municipality
  - Jiading Central Hospital, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Taizhou Hospital of Zhejiang Province - Main, Taizhou, Zhejiang
- Colombia (2):
  - Clinica de la Costa S.A.S. - PPDS, Barranquilla, Atlántico
  - Healthy Medical Center S.A.S., Zipaquirá, Cundinamarca
- Croatia (4):
  - Klinicki bolnicki centar Sestre Milosrdnice - Vinogradska cesta 29, Zagreb, City of Zagreb
  - Polyclinic Bonifarm, Zagreb, City of Zagreb
  - Clinical Hospital Center Rijeka, Rijeka
  - Special Hospital Medico, Rijeka
- Institut klinicke a experimentalni mediciny, Prague, Praha, Hlavní Mesto, Czechia
- France (13):
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg, Bas-Rhin
  - CHU de Besançon, Besançon, Dobus
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux, Gironde
  - CHU de Reims - Hôpital Maison Blanche, Reims, Grand Est
  - GHRMSA - Hôpital Emile Muller, Mulhouse, Haut-Rhin
  - Hopital Foch, Suresnes, Hauts-de-Seine
  - CHRU d'Orleans- Hôpital de La Source, Orléans, Loiret
  - CHU de Nîmes - Hopital Universitaire Caremeau, Nîmes Cédex 9, Occitanie
  - AP-HP - Hôpital Henri Mondor, Créteil, Val-de-Marne
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon, Vendée
  - CHU Amiens Picardie - Site Sud, Dreuil-lès-Amiens
  - AP-HP - Hôpital Saint-Louis, Paris
  - AP-HP - Hopital Tenon, Paris
- Germany (3):
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt, Apotheke Haus 19, Frankfurt am Main, Hesse
  - Charité - Universitätsmedizin Berlin, Berlin
- Greece (3):
  - General Hospital of Athens ''G. Gennimatas'', Athens, Attica
  - Laiko General Hospital of Athens, Athens, Attica
  - General Hospital of Heraklion Venizeleio, Heraklion, Irakleio
- India (13):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Nizams Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - All India Institute of Medical Sciences ( AIIMS ) - Raipur, Raipur, Chhattisgarh
  - Zydus Hospital, Ahmedabad, Gujarat
  - M.S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Trivandrum Medical College Hospital, Trivandrum, Kerala
  - Seth G S Medical College and K E M Hospital, Mumbai, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Max Super Speciality Hospital - Saket, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - King George Medical University, Lucknow, Uttar Pradesh
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West Bengal
- Italy (5):
  - AUSL Piacenza - Ospedale Guglielmo da Saliceto, Piacenza, Emilia-Romagna
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - Ospedale di Cattinara, Trieste, Friuli Venezia Giulia
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia, Lombardy
  - Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò, Ranica, Lombardy
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara, Piedmont
- Japan (20):
  - Fujita Health University Hospital, Toyoake-shi, Aiti
  - National Hospital Organization Chiba Medical Center Chibahigashi National Hospital, Chiba, Chiba
  - Juntendo University Urayasu Hospital, Urayasu-Shi, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi, Hukuoka
  - Fukushima Medical University Hospital, Fukushima, Hukusima
  - Toranomon Hospital Kajigaya, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyôto
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Hamamatsu University Hospital, Hamamatsu, Sizouka
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Showa Medical University Hospital, Shinagawa-ku, Tokyo
  - Ikeda Municipal Hospital, Ikeda-shi, Ôsaka
  - Osaka University Hospital, Suita-shi, Ôsaka
- Malaysia (3):
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun, Perak, Pahang
  - University Malaya Medical Centre, Lembah Pantai, WilayahPersekutuan KualaLumpur
- Norzel Medical and Diagnostic Clinic Foundation Corp., Cebu City, Cebu, Philippines
- Poland (4):
  - MCM Krakow - PRATIA - PPDS, Krakow, Lesser Poland Voivodeship
  - SCM Clinic - Prywatny Szpital Specjalistyczny, Krakow, Lesser Poland Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
- Portugal (7):
  - ULS de Lisboa Ocidental, EPE - Hospital Santa Cruz, Carnaxide, Lisbon District
  - ULS de Gaia/Espinho, EPE - Unidade I, Vila Nova de Gaia, Lisbon District
  - ULS da Região de Aveiro, EPE - Hospital Infante D. Pedro, Aveiro
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - ULS da Região de Leiria, EPE - Hospital de Santo André, Leiria
  - ULS da Arrábida, EPE - Hospital de São Bernardo, Setúbal
- FDI Clinical Research, San Juan, Puerto Rico
- South Korea (9):
  - Pusan National University Hospital, Busan, Gwangyeogsi
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Ajou University Hospital, Suwon, Gyeonggido
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospital, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (12):
  - Fundacio Puigvert, Viladecans, Barcelona
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital General San Pedro de Alcantara, Cáceres
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (8):
  - National Cheng Kung University Hospital, Dawan, Taiwan, Province of China
  - Far Eastern Memorial Hospital, New Taipei City, Taiwan, Province of China
  - China Medical University Hospital - PPDS, Taichung, Taiwan, Province of China
  - Mackay Memorial Hospital-Taipei branch, Taipei, Taiwan, Province of China
  - Taipei Municipal Wanfang Hospital, Taipei, Taiwan, Province of China
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan, Province of China
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
- Turkey (Türkiye) (2):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
- United Kingdom (3):
  - Royal Preston Hospital - NWCRN- PPDS, Preston, Lancashire
  - Leicester General Hospital, Leicester, Leicestershire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/